CLINICAL TRIAL: NCT05418894
Title: Mapping and Modulating the Spatiotemporal Dynamics of Socio-Affective Processing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kelly Bijanki, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5R01MH127006-02 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Treatment Resistant Depression; Epilepsy
Keywords: Deep Brain Stimulation; Neuromodulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EMU (No Intervention): Patient's behavioral and neural activity via computer tasks and questionnaires are monitored in the Epilepsy Monitoring Unit
- TRD (Experimental)
  Interventions: Device: Device: Directional Deep Brain Stimulation

INTERVENTIONS:
Device: Device: Directional Deep Brain Stimulation — Boston Scientific Vercise DBS leads and 16-channel implanted pulse generators (IPGs) will be implanted to control the shape and size of stimulation
  Arms: TRD

SUMMARY:
The overall goal of this study is to map the spatiotemporal dynamics of social affective processing and to examine selective modulation of these dynamics in humans undergoing invasive intracranial monitoring for treatment-resistant epilepsy and depression. Pursuing this signal from a novel platform with invasive intracranial recording electrodes provides much-needed spatial and temporal resolution to characterize the neural dynamics of socio-affective processing. The investigators will leverage first-in-human intracranial neural recording opportunities created by a novel therapeutic platform termed "stereotactic electroencephalography-informed deep brain stimulation" (stereo-EEG-informed DBS), as well as the powerful platform of intracranial stereotactic recording and stimulation in patients undergoing epilepsy surgical evaluation at Baylor College of Medicine. The sEEG-informed DBS trial provides unique opportunities for intracranial recording of affect-relevant network regions in patients with treatment-resistant depression (TRD). Recordings in identical regions in epilepsy patients who themselves often demonstrate mild-moderate depressive symptoms will provide a wide dynamic range across the symptom spectrum. To provide critical data on the spatiotemporal dynamics of socio-affective processing the investigators will leverage these two human intracranial recording and stimulation cohorts to study the precise structural, functional, and causal properties of the affective salience network. Greater understanding of the social processing circuitry mediated by the affective salience network may be used to drive therapeutic innovation, pioneering a new paradigm that improves socio-emotional function across a wide variety of neuropsychiatric conditions. The results from this proposal have the potential to improve the lives of patients with dysfunction in social affective processing, with implications for a wide range of neuropsychiatric diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-pregnant) between ages 22 and 70;
2. DSM-5 diagnosis (assessed by Structured Clinical Interview for DSM-5 Axis I disorders SCID-5) of major depression disorder (MDD) as the primary diagnosis. A current major depressive episode (MDE), recurrent or single episode with first episode before age 60, secondary to nonpsychotic unipolar major depressive disorder;
3. Chronic illness with current MDE ≥24 months duration and/or recurrent illness with at least a total of 2 lifetime episodes (including current episode >12 months);
4. Treatment resistance (defined by criteria on the Antidepressant Treatment History Form ATHF): Failure (i.e. persistence of the major depressive episode) to respond to a minimum of four adequate depression treatments from at least two different treatment categories (e.g. SSRIs, SNRIs, TCAs, other antidepressants, lithium-addition, irreversible MAOIs, antidepressant augmentation with an atypical antipsychotic medication);
5. Previous trial of Electroconvulsive Therapy (ECT) (lifetime): either did not respond, relapsed, poorly tolerated or refused. If refused, will discuss reasons and ensure subject understands relative risks of ECT versus DBS. We will try to enrich sample with patients who had previously shown response to ECT (or another intervention) that was partial or un-sustained;
6. Symptom severity for Screening: Hamilton Depression Rating Scale-17 item (HDRS17)

   ≥20;
7. The HDRS17 must remain greater than or equal to 20 on two separate assessments (at initial screening and 1 week before surgery), over a 1-month period;
8. Symptom severity for Outcome: Montgomery Asberg Rating Scale (MADRS) ≥27 to be met at assessment one-week pre-op;
9. Lifetime exposure to minimal 6 weeks of psychotherapy without sustained response;
10. Must have a brain MRI within 3 months of enrollment that is "normal", according to the radiology report, or does not reveal any findings that in the opinion of the Investigator preclude participation in the study;
11. Stable antidepressant medication regimen for the month preceding surgery;
12. Modified mini-mental state examination (MMSE) score ≥ 24;
13. Normal thyroid stimulating hormone (TSH) level within 12 months of study entry;
14. The patient does not have any medical or physical conditions which, in the opinion of the Investigator, make it unlikely the patient will be able to participate for the duration of the study;
15. Able and willing to give informed consent and agree to attend regular clinic visits for at least 12 months following surgery;
16. Must have a treating psychiatrist, a family member, significant other/living partner, a caregiver, or a person known by the subject present at the Screening visit for the discussion about the study before co-signing the informed consent form;
17. Willingness to sign Treatment Contract;
18. Agrees to be followed at regular intervals by a licensed psychiatrist and to provide written permission allowing any and all forms of communication between the research team and the subject's healthcare providers, for the entirety of the study;
19. Both male and female patients who undergo placement of intracranial electrodes for clinical characterization of epilepsy.

Exclusion Criteria:

1. DSM-5 Axis I Disorders: any lifetime history of psychotic disorder (e.g., schizophrenia, schizoaffective disorder);
2. Bipolar disorder with rapid cycling and history of manic episode requiring hospitalization within the past 5 years;
3. Clinically significant Cluster A or B personality disorder;
4. Alcohol or substance use disorder within 6 months, excluding nicotine;
5. Urine drug test positive for illicit drugs;
6. Any evidence or indication of suicidal intent, suicidal attempt, or suicidal behavior, including but not limited to the C-SSRS score, within the past one year;
7. Neurological/Medical condition that makes the patient, in the opinion of the surgeon, a poor surgical candidate (e.g., progressive neurodegenerative disorder, significant cardiopulmonary disorder, need for chronic anticoagulation);
8. Any history of seizure disorder, hemorrhagic stroke, or has high risk of seizure (history of congenital brain malformation, history of brain injury, neuro-developmental disorder, currently taking medication that is known to lower seizure threshold, or other factors that predispose seizures);
9. Any medical contraindication to surgery such as infection;
10. Coagulopathy: Bleeding propensity and/or one of the following: INR > 1.5; prolonged activated partial thromboplastin time (aPTT) ≥ 45 sec; platelet count < 100×103/uL;
11. A blood pressure of ≥ 180/110 mmHg at a single visit and evidence of cardiovascular disease (CVD);
12. Participation in another drug, device, or biological trial within 90 days;
13. Current implanted stimulation devices including cardiac pacemakers, defibrillators, and neurostimulators including spinal cord stimulators and deep brain stimulators;
14. Pregnant or has plans to become pregnant in the next 24 months;
15. Anticipated need for MRI;
16. Need for Diathermy;
17. Chronic use of anticoagulant or anti-platelet agents that cannot be safely stopped for a sufficient duration (minimum 2.5 weeks) in the peri-operative period.
18. Any Psychiatric/Neurological/Medical condition that makes the subject, in the opinion of the Investigator, a poor candidate.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of streamlines connecting between intracranial stimulation volume and recording volumes. | up to 8 weeks
  To characterize structural connectivity using diffusion-weighted neuroimaging, we will calculate the outcome measures of the number of streamlines connecting target points.
Evoked potentials arising from stimulation. | up to 8 weeks
  To characterize short latency mono- or oligo-synaptic connections of the stimulation volumes to sEEG recording positions using the single pulse-evoked potentials (PEP) technique, the outcome measure will be the number of evoked potentials arising from applied stimulation.

SECONDARY OUTCOMES:
Spectral band power during mood-relevant cognitive task. | up to 12 weeks
  We will characterize the electrophysiological function of the affective salience network via the outcome measure of local field potential recordings in terms of power spectral density during mood-relevant cognitive function.
Spectral band power following applied stimulation. | up to 8 weeks
  We will measure the outcome measure of local field potential power spectral density following the application of research stimulation.
Match score between spectral band power matrix of desired state and stimulation-evoked state. | up to 12 weeks
  We will implement a process of template-matching to align stimulation-evoked neural activity patterns with "desirable" neural state signatures, including natural and induced positive mood states, using spatiotemporal correlation matrix decomposition and machine learning dimensionality reduction. The outcome measure will be the degree of correlational match between desired state and various evoked states following stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States